CLINICAL TRIAL: NCT04929262
Title: Increasing Parent Demand for Evidence-Based Practices to Treat Youth Anxiety: The Effect of Parent Key Opinion Leaders
Brief Title: Parent Key Opinion Leaders to Increase Demand of Effective Treatments for Youth Anxiety
Acronym: Project CHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Illinois at Chicago (Other); Brown University (Other); Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 26871; 1F31MH124346-01 (NIH)
Record Dates: First submitted 2021-06-03; First posted 2021-06-18 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Anxiety Disorders
Keywords: dissemination; key opinion leader; direct-to-consumer marketing; healthcare utilization; evidence-based practice; youth anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Researcher-Only (Active Comparator): The researcher-facilitated presentation, led by two clinical psychology graduate students, will be the same for all schools.
  Interventions: Behavioral: Supporting Anxious Youth: Strategies for Caregivers
- Key Opinion Leader (Experimental): The key opinion leader (KOL) co-facilitated presentations will include the same core principles as the researcher-facilitated presentation but may vary by school in terms of specific examples and content emphasized based on KOL feedback. A caregiver KOL from the local community (selected by the parent teacher association or a similar group) will co-facilitate the presentation with a clinical psychology graduate researcher.
  Interventions: Behavioral: Supporting Anxious Youth: Strategies for Caregivers

INTERVENTIONS:
Behavioral: Supporting Anxious Youth: Strategies for Caregivers — The outreach presentation will last 75 minutes with an additional 15 minutes for caregiver questions. The presentations will occur in the evening via Zoom. The presentation will include information about identifying anxiety disorders, strategies for caregivers to help their youth with anxiety, evidence-based practices to treat youth anxiety, and strategies for finding a therapist who uses cognitive behavior therapy with exposures. The text on the presentations is written at a 5.3 grade reading level. Presentations will incorporate stigma reduction strategies, such as education to dispel myths, and behavioral decision-making tools to elicit hope, empowerment, and motivation.

SUMMARY:
Despite research identifying effective treatments for youth anxiety, parents (and other primary caregivers) are unaware that some treatments are more effective than others. This study investigates whether having a local parent key opinion leader co-facilitate an educational outreach presentation on effective treatment for youth anxiety will increase parent demand for evidence-based practices (EBPs). It is hypothesized that participants who receive a presentation co-presented by a key opinion leader will be more likely to have sought cognitive behavioral therapy for their child at the three-month follow up, relative to participants who receive a presentation presented by two researchers.

DETAILED DESCRIPTION:
Anxiety disorders are common among adults and youth and, when left untreated, are associated with several long-term negative sequelae. Although research has identified a number of EBPs for treating youth anxiety (in particular, cognitive behavioral therapy [CBT] with exposures) and despite large-scale implementation efforts, few youth receive EBPs. Direct-to-consumer marketing offers a different approach to increase provider uptake of EBPs by increasing parent demand for EBPs. Direct-to-consumer initiatives are especially important given patient-barriers that prevent youth from receiving treatment, including lack of parental knowledge of EBPs and stigma associated with mental health treatment. Although parent preferences for receiving information about EBPs vary based on demographic factors and individual experiences, research has not investigated methods of tailoring direct-to- consumer efforts to local contexts. Involving a local parent key opinion leader (KOL) to tailor direct-to- consumer initiatives to local contexts may be an effective strategy to increase parent demand for EBPs. KOLs are credible and trustworthy members of a local community who can use their social influence to disseminate information and validate messages about EBPs. Research indicates that KOLs improve health promotion campaigns, but KOLs have not been studied in the context of increasing parent demand for EBPs. The project will examine the role of KOL participation in conducting outreach presentations to increase parent desire to seek CBT for their youth's anxiety. Parent attendees (or primary caregivers; N = 180) will be cluster-randomized by school to one of two different approaches for presentations on EBPs for youth anxiety (90 parents per condition). Both approaches will include community outreach presentations providing information about youth anxiety, effective treatments for youth anxiety, and seeking CBT for youths. The researcher-only condition will be co-facilitated by two researchers. In the KOL condition, a parent KOL from each local community will be involved in tailoring the content of the presentation to the context of the community, co-facilitating the presentation with a researcher, and endorsing strategies in the presentation that they have found to be helpful. The parent-teacher association (or a similar group of parents) from each school will nominate a parent who is well-known and well-respected within their community as the KOL. Parent attendees for both conditions will be recruited by contacting school mental health workers/other school administrators, who will advertise the presentations via their school email list and fliers sent home with children. Parent attendees will complete measures assessing their knowledge of, attitudes towards, and intention to seek CBT pre- and post- presentation, and they will indicate whether they sought CBT for their youth at a three-month follow-up. This study will use a mixed methods approach (integrating quantitative and qualitative methods) to test the effect of KOLs on increasing caregiver demand for CBT for youth anxiety. Primary aims test the relative effects of researcher-only and KOL conditions on changing caregivers' intention to seek CBT for their youth, and actual CBT seeking at three-month follow up. Secondary aims examine (1) the relative effects of researcher-only and KOL conditions on changing caregivers' perceived subjective norms about seeking CBT, attitudes about CBT, stigma about mental illness, and knowledge of how to seek EBPs; and (2) how KOLs affect participants' impression of the researcher presenter. This study will provide future direct-to-consumer efforts with evidence about effective strategies to increase parent demand for EBPs, which in turn will enable parents to seek the best care for their child.

ELIGIBILITY:
Inclusion Criteria:

* Be least 18 years of age
* Be fluent in English
* Be the primary caregiver of a youth aged 5 to 18 years
* Have a child at one of the schools offering a presentation

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Kendall, Ph.D., Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crane ME, Atkins MS, Becker SJ, Purtle J, Olino TM, Kendall PC. The effect of caregiver key opinion leaders on increasing caregiver demand for evidence-based practices to treat youth anxiety: protocol for a randomized control trial. Implement Sci Commun. 2021 Sep 23;2(1):107. doi: 10.1186/s43058-021-00213-x. PMID 34556182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Elementary, middle, and high schools located within a 1.5-hour drive of Philadelphia were recruited by emailing their school mental health workers/other school administrators. School administrators advertised presentations as they advertise other school events (e.g., email list, Facebook groups).
Units Other Than Participants: School
Period: Pre-Presentation Questionnaires
Arm/Group | Researcher-Only | Key Opinion Leader
Started | 152; 14 School | 131; 13 School
Completed | 112; 13 School | 97; 12 School
Not Completed | 40; 1 School | 34; 1 School
Period: Attended Presentation
Arm/Group | Researcher-Only | Key Opinion Leader
Started | 112; 13 School | 97; 12 School
Completed | 57; 13 School | 52; 12 School
Not Completed | 55; 0 School | 45; 0 School
Period: Post-Presentation Questionnaires
Arm/Group | Researcher-Only | Key Opinion Leader
Started | 57; 13 School | 52; 12 School
Completed | 49; 13 School | 47; 12 School
Not Completed | 8; 0 School | 5; 0 School
Period: 3 Month Follow-Up Questionnaires
Arm/Group | Researcher-Only | Key Opinion Leader
Started | 57; 13 School | 52; 12 School
Completed | 39; 13 School | 36; 12 School
Not Completed | 18; 0 School | 16; 0 School

BASELINE CHARACTERISTICS:
Population: Number of participants who completed the demographic questionnaire
Groups:
- Total: Total of all reporting groups
Arm/Group | Researcher-Only | Key Opinion Leader | Total
Number analyzed (Participants) | 113 | 97 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant chose not to disclose their age
  years
    number analyzed (Participants) | 112 | 97 | 209
    (all) | 40.31 (7.19) | 41.06 (6.29) | 40.66 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant chose not to disclose their sex
  Participants
    number analyzed (Participants) | 113 | 96 | 209
    Female | 104 | 89 | 193
    Male | 9 | 7 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 21 | 33
  Not Hispanic or Latino | 99 | 74 | 173
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Category options were not mutually exclusive; respondents could select multiple races/ethnicities
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 3 | 3 | 6
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 23 | 16 | 39
    White | 80 | 60 | 140
    More than one race | 2 | 3 | 5
    Unknown or Not Reported | 5 | 14 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre-Presentation to Post-Presentation in Treatment Seeking Evaluation - Intention to Seek Cognitive Behavioral Therapy
Description: Participants rate how likely they are to seek a therapist who uses exposure therapy for their child in the next three months on a scale ranging from 1 (very unlikely) to 5 (very likely).
Time Frame: pre-presentation; post-presentation (within 1 week after the presentation)
Population: The overall number of participants analyzed is greater than the number of participants who completed the pre-presentation questionnaires because some participants completed this measure, but not the entire pre-presentation questionnaire battery. The data reported includes responses from all participants who completed the measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Researcher-Only | Key Opinion Leader
Number analyzed (Participants) | 114 | 98
score on a scale
  Pre-presentation | 3.23 (1.18) | 3.02 (1.22)
  Post-presentation: number analyzed (Participants) | 49 | 47
  Post-presentation | 3.67 (1.20) | 3.79 (1.18)

2. Primary Outcome: Number of Participants Who Sought Cognitive Behavioral Therapy as Assessed by Treatment Seeking Evaluation - Actual Cognitive Behavioral Therapy Seeking
Description: Participants indicate whether they sought exposure therapy for their child since the presentation. Participants were first ask if they sought therapy for their child. If yes, they were asked if they sought exposure therapy for their child (options were yes, no, unsure). The count provided is the number of participants that responded "yes" they sought exposure therapy for their child.
Time Frame: 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Researcher-Only | Key Opinion Leader
Number analyzed (Participants) | 39 | 36
Participants | 3 | 3

3. Secondary Outcome: Change From Pre-Presentation to Post-Presentation in Parent Engagement in Evidence-Based Services Questionnaire, Knowledge Subscale
Description: The Parent Engagement in Evidence-Based Services Questionnaire, Knowledge subscale assesses caregiver perceived understanding of how to seek evidence-based practice. Participants rate five items on a ranging from 1 (strongly disagree) to 5 (strongly agree). Items are averaged to create the Parent Engagement in Evidence-Based Services Questionnaire, Knowledge subscale (subscale range = 1-5); higher scores indicate higher levels of perceived knowledge about seeking evidence-based practice.
Time Frame: pre-presentation; post-presentation (within 1 week after the presentation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Researcher-Only | Key Opinion Leader
Number analyzed (Participants) | 129 | 109
score on a scale
  Pre-Presentation | 3.01 (0.74) | 3.06 (0.74)
  Post-Presentation: number analyzed (Participants) | 50 | 48
  Post-Presentation | 3.56 (0.61) | 3.70 (0.72)

4. Secondary Outcome: Change From Pre-Presentation to Post-Presentation in Therapy Subjective Norms Questionnaire
Description: The Therapy Subjective Norms Questionnaire is a six-item measure of caregiver perception of subjective norms for seeking cognitive behavioral therapy. Items are rated on a scale ranging from 1 (strongly disagree) to 7 (strongly agree). Items are summed to create a total score (range = 6 - 42); higher scores indicate more positive subjective norms about seeking therapy.
Time Frame: pre-presentation; post-presentation (within 1 week after the presentation)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Researcher-Only | Key Opinion Leader
Number analyzed (Participants) | 124 | 104
units on a scale
  Pre-Presentation | 32.60 (6.98) | 31.36 (7.40)
  Post-Presentation: number analyzed (Participants) | 50 | 47
  Post-Presentation | 34.28 (6.71) | 33.81 (6.35)

5. Secondary Outcome: Change From Pre-Presentation to Post-Presentation in Caregiver Attitudes About Cognitive Behavioral Therapy
Description: The Caregiver Attitudes about Cognitive Behavioral Therapy includes 18 strategies used in cognitive behavioral therapy for youth anxiety. Participants rate how helpful they believe each strategy would be for treating their child on a five-point scale ranging from 1 (very unhelpful) to 5 (very helpful). Items are summed to create a total score (range = 18 - 90); higher scores indicate more favorable attitudes.
Time Frame: pre-presentation; post-presentation (within 1 week after the presentation)
Population: The number of participants analyzed is greater than the number of participants who completed the pre-presentation questionnaires because some participants completed this measure, but not the entire pre-presentation questionnaire battery. The data reported includes responses from all participants who completed the measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Researcher-Only | Key Opinion Leader
Number analyzed (Participants) | 114 | 99
units on a scale
  Pre-Presentation | 80.35 (11.94) | 79.04 (8.63)
  Post-Presentation: number analyzed (Participants) | 49 | 47
  Post-Presentation | 82.98 (8.24) | 81.13 (7.52)

6. Secondary Outcome: Change From Pre-Presentation to Post-Presentation in Parents' Internalized Stigma of Mental Illness Scale
Description: The Parents' Internalized Stigma of Mental Illness Scale (PISMIS) assesses caregiver perception of internalized stigma for having a youth with a mental illness (Zisman-Ilani et al., 2013). Participants rate 10 statements on a scale ranging from 1 (strongly disagree) to 4 (strongly agree); some items are reverse scored. Items are summed to create a total score (range = 10-40); higher scores indicate higher levels of family stigma.
Time Frame: pre-presentation; post-presentation (within 1 week after the presentation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Researcher-Only | Key Opinion Leader
Number analyzed (Participants) | 137 | 112
units on a scale
  Pre-Presentation | 15.07 (4.26) | 15.01 (5.00)
  Post-Presentation: number analyzed (Participants) | 50 | 48
  Post-Presentation | 14.90 (4.30) | 14.60 (5.90)

7. Other Pre Specified Outcome: Change From Pre-Presentation to Post-Presentation and to 3-Month Follow-Up in Barriers to Seeking Treatment
Description: The Barriers to Seeking Treatment questionnaire asks participants to indicate whether they agree with 21 potential barriers to treatment (yes/no). A count of the total number of barriers will be used in analyses.
Time Frame: pre-presentation; post-presentation (within 1 week after the presentation)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change From Pre-Presentation to 3-Month Follow-Up in Barriers to Seeking Treatment
Description: as for outcome 7
Time Frame: pre-presentation; 3-month follow-up
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Client Satisfaction Questionnaire
Description: The Client Satisfaction Questionnaire assesses participants' satisfaction with the presentation. Items are rated on scale ranging from 1 to 4. Items are summed; higher composite scores indicate greater program satisfaction.
Time Frame: post-presentation (within 1 week after the presentation)
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Relatability Evaluation
Description: The Relatability Evaluation will be used to evaluate participants' impression of the presenter. Participants will rate each presenter (scale ranging from 1 to 5) on 10 items associated with aspects of key opinion leaders: relatable, likeable, similar, think similarly, similar beliefs, credible, trustworthy, understanding of the local community, familiar, and friendship. Items are summed; higher composite scores indicate that the presenter is more relatable.
Time Frame: post-presentation (within 1 week after the presentation)
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Brief Revised Child Anxiety and Depression Scale-Parent Version
Description: The total anxiety scale (15 items) from the Brief Revised Child Anxiety and Depression Scale-Parent Version will be used to assess youth anxiety (Ebesutani et al., 2017). Participants rate items on a scale from 0 (never) to 3 (always). Items are summed; higher scores indicate higher levels of anxiety.
Time Frame: pre-presentation
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Demographics
Description: A demographics questionnaire will assess caregiver and youth age, gender, race, ethnicity, and nativity; caregiver level of education, income, and religion; and youth health insurance status.
Time Frame: pre-presentation
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Content Checklist
Description: A content checklist will assess the core components of the presentation, as well as presenter and audience member self-disclosure about experiencing receiving therapy for themselves or their child (yes/no). Self-disclosure will be considered to have been made if either the presenter or an audience member self-discloses about their experiences.
Time Frame: during the 1.5 hour presentation
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Qualitative Interview
Description: A qualitative interview will ask participants about the following topics: (1) their perception of presenters; (2) ways in which the presenters affected their decision to seek treatment; (3) factors they considered when seeking treatment; (4) strategies they have used from the presentation; (5) their perception of exposure therapy; and (6) general ways that the mental health system could be improved to improve access to therapy.
Time Frame: 3-month follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Description: During the course of the intervention and follow up period.
Arm/Group | Researcher-Only | Key Opinion Leader
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/131
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/131
Other Adverse Events (participants affected / at risk) | 0/152 | 0/131

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT04929262/Prot_SAP_002.pdf
  • Informed Consent Form (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT04929262/ICF_003.pdf